CLINICAL TRIAL: NCT01193491
Title: A Phase 1 Open-Label, Dose Escalation Study Evaluating the Safety and Tolerability of IPI-493 in Patients Experiencing Advanced Hematologic Malignancies With Client Proteins of Hsp90
Brief Title: Dose Escalation of IPI-493 in Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug exposure of retaspimycin HCl was superior to IPI-493, Infinity will focus on Retaspimycin HCL
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-493-02
Record Dates: First submitted 2010-06-28; First posted 2010-09-02 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Hematologic Malignancies
Keywords: Phase 1; AML; CML; MPD; Client Proteins; Hsp90
MeSH Terms: conditions — Hematologic Neoplasms | interventions — tanespimycin; HSP90 Heat-Shock Proteins; geldanamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-493 (Experimental)
  Interventions: Drug: IPI-493

INTERVENTIONS:
Drug: IPI-493 — Capsules, ascending dose, multiple schedules
  Other Names: HSP-90; Geldanamycin

SUMMARY:
The purpose of this study is to evaluate the safety, determine the maximum tolerated dose (MTD) and schedule of IPI-493 in patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* >/=18 years old
* ECOG 0-1
* confirmed hematological malignancy
* refractory to available therapy or for which no therapy is available
* adequate hepatic, renal function

Exclusion Criteria:

* active CNS malignancy
* prolonged QT interval
* significant GI/liver disease
* other serious concurrent illness or medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety Endpoints | 1 year
  Safety Endpoints
  * The incidence of reported adverse events (AEs), serious adverse events (SAEs), concomitant medication use, laboratory test results, electrocardiogram (ECG) results, Eastern Cooperative Oncology Group (ECOG) performance status results, and vital sign results
  * Maximum tolerated dose, defined as the dose level below the dose at which ≥33% of patients experience a dose limiting toxicity (DLT) Pharmacodynamic Endpoints

SECONDARY OUTCOMES:
Evaluation of Efficacy Endpoints | 1 year
Evaluation of Efficacy Endpoints | 1 year
  * Hematologic disease-specific outcomes for response including but not limited to complete hematologic response (CHR) and partial hematologic response (PHR)
  * Plasma concentrations of IPI-493 (and IPI-493 metabolites, if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, M.D., Study Director — Infinity Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Johns Hopkins Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Weill Cornell Cancer Center, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas